CLINICAL TRIAL: NCT06285006
Title: Predictors of Success and Relapse After Desmopressin Monotherapy for Monosymptomatic Nocturnal Enuresis
Brief Title: Desmopressin Monotherapy for Monosymptomatic Nocturnal Enuresis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hosny Mohamed Ahmed Elmasry, Professor, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MScAZASTPED025/23/202/12/2021
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Nocturnal Enuresis
Keywords: Nocturnal enuresis; Desmopressin; Monotherapy
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Desmopressin (Experimental): Desmopressin is a synthetic analogue of ADH released by the posterior pituitary gland that reduces urine production by increasing water reabsorption by the collecting tubules.
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Desmopressin is a synthetic analogue of ADH released by the posterior pituitary gland that reduces urine production by increasing water reabsorption by the collecting tubules.

SUMMARY:
Nocturnal Enuresis (NE) is defined as the involuntary passage of urine during sleep past the age of usual control, which is considered a developmental age of 5 to 7 years.

NE is a common problem that causes distress to both children and their families. It has an adverse impact on behavior and social life, affects self-esteem, and can result in poor emotional well-being. In Egypt, the prevalence of NE in primary school children is about 15.4%. The family history was seen to have had a markedly significant impact on the occurrence of NE in the studied children. The mainstay of treatment is urotherapy with information and psychoeducation about normal lower urinary tract function, the underlying cause of MNE, disturbed bladder dysfunction in the child with NMNE, and instructions about therapeutic strategies. Alarm therapy and desmopressin are effective in randomized trials. Children with NMNE first need treatment of the underlying daytime functional bladder problem before treatment of nocturnal enuresis.

ELIGIBILITY:
Inclusion Criteria:

* School age group (from 7 to 14 years)
* Primary monosymptomatic nocturnal enuresis

Exclusion Criteria:

Patients with one or more of the following will be excluded from the study.

* Diurnal enuresis
* Urinary tract infection within the preceding 3 months
* Diabetes mellitus
* History of renal disease, hypertension or genitourinary abnormality, neurological disease, or psychological disease.
* Post-micturition residual urine >1/3 expected bladder capacity.
* Each patient will be subjected to the following.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-12 (Estimated)

PRIMARY OUTCOMES:
The number of episodes per week after desmopressin treatment | After the end of the treatment for one month.
  Patients will be evaluate by no. of episodes per week after desmopressin treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No